CLINICAL TRIAL: NCT04163289
Title: Preventing Immune-Related Adverse Events in Renal Cell Carcinoma Patients Treated With Combination Immunotherapy Using Fecal Microbiota Transplantation
Brief Title: Preventing Toxicity in Renal Cancer Patients Treated With Immunotherapy Using Fecal Microbiota Transplantation
Acronym: PERFORM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERFORM Renal
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Fecal microbiota transplantation combined with approved standard of care treatment with nivolumab and ipilimumab.
  Interventions: Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Fecal microbiota transplantation is the process of administering stool samples derived from healthy donors, which have been processed and prepared into capsules. Capsules will be taken 7 days or more prior to the first treatment with nivolumab and ipilimumab, and 1 to 3 days prior to the next 2 treatments with nivolumab and ipilimumab.

SUMMARY:
Cancer immunotherapy has been largely adopted in oncology patient management in the last decade. The deep and long responses to immunotherapy have accelerated the approval of these drugs across multiple disease sites. However, these agents can also be toxic to patients, meaning, the patient will have to discontinue treatment and outcomes could be negatively affected. Recently, a combination of two immunotherapy drugs, ipilimumab and nivolumab (ipi/nivo), has been approved for the treatment of intermediate and poor-risk renal cell carcinoma (RCC) patients. This powerful combination provides survival benefit, however, it can also be highly toxic leading to discontinuation of this treatment.

There has been some evidence that these otherwise toxic drugs can be better tolerated by altering the composition of the patients gut bacteria to create a more diverse and healthy microbiome. The current study will involve Fecal Microbiota Transplantation (FMT) before the start of the immunotherapy combination, and during the first two cycles of ipilimumab treatment (the more toxic agent) as supportive therapy to prevent toxicity associated with the ipi/nivo combination.

The goal of this project is to study the safety of such FMT combination treatment and reduce occurrence of immune-related toxicities in patients, allowing them to continue their cancer treatments in the hopes of a better outcome. The investigators will also be looking at changes in the immune populations, microbiome profile of patients, response to treatment, and patient survival as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) renal cell carcinoma
* Intermediate or poor risk RCC as defined by International Metastatic RCC Database Consortium (IMDC criteria, Heng et al 2009):

  * Karnofsky performance status (KPS) < 80%
  * Less than 1 year form initial RCC diagnosis (including original localized disease if applicable) to systemic treatment
  * Hemoglobin < lower limit of normal (LLN)
  * Corrected calcium > 10 mg/dL
  * Absolute neutrophil count (ANC) > upper limit of normal (ULN)
  * Platelet count > ULN
* Age ≥ 18 years.
* Karnofsky Performance Status (KPS) ≥70%
* Evaluable disease determined by the Investigator
* Ability to ingest capsules
* Able to provide written informed consent
* Understand non-infectious risks associated with FMT administration and that the long term data regarding safety risks of FMT are lacking
* Recovery to baseline or ≤ Grade 1 CTCAE v 4.0 from toxicities related to any prior treatments, unless AEs are clinically non-significant
* Adequate organ and marrow function, based upon meeting all the following laboratory parameters:

  1. Absolute neutrophil count (ANC) ≥ 1500/μL (≥ 1.5 x 109/L) without granulocyte colony-stimulating factor support within 4 weeks before screening laboratory sample collection.
  2. White blood cell count ≥ 2000/μL (≥ 2.0 x 109/L)
  3. Platelets ≥ 100,000/μL (≥ 100 x 109/L) without transfusion within 4 weeks before screening laboratory sample collection.
  4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L) without transfusion within 4 weeks before screening laboratory sample collection.
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
  6. Total bilirubin ≤ 1.5 × ULN (with the exception that total bilirubin for subjects with Gilbert's disease ≤ 3 × ULN).
  7. Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft-Gault equation (see for Cockcroft-Gault formula).
  8. Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol), or 24-h urine protein ≤ 1 g

Exclusion Criteria:

* Prior systemic therapy for unresectable locally advanced or metastatic RCC including investigational agents.
* Radiation therapy for bone metastasis within 2 weeks, or any other radiation therapy within 4 weeks prior to study entry. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible for the study.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with signing the informed consent through 6 months after FMT.
* Diagnosis of immunodeficiency (e.g. HIV, transplantation)
* Receiving systemic steroid therapy (>10mg prednisone daily or equivalent) or any other form of immunosuppressive therapy prior to trial treatment. Adrenal replacement steroids doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic steroids for allergic situations (e.g. contrast allergy) is also permitted. Patients who require inhaled, intranasal, intra-articular, or topical steroids are allowed. Intermittent use of bronchodilators or local steroid injections are not excluded from the study
* Ongoing use of antibiotics or previous use of antibiotics in the last two weeks prior to the initial FMT procedure
* Presence of a chronic intestinal disease (e.g. Celiac, malabsorption, colonic tumor)
* Presence of absolute contra-indications to FMT administration

  * Toxic megacolon
  * Severe dietary allergies (e.g. shellfish, nuts, seafood)
  * Inflammatory bowel disease
* Expected to require any other form of systemic or localized anti-neoplastic therapy while on study. Treatment with either bisphosphonate or denosumab for bone metastatic disease is allowed
* Known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years

  o NOTE: This time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
* Active central nervous system (CNS) metastases and/or leptomeningeal involvement, unless treated with radiotherapy and/or radiosurgery with stable disease for at least 4 weeks prior to study entry after radiotherapy or at least 8 weeks prior to study entry after major surgery
* Active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.

  o Patients with vitiligo, type I diabetes, resolved childhood asthma/atopy are exceptions to this rule
* A history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Serious concomitant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders

  o This includes HIV or AIDS-related illness, or active HBV and HCV
* Active infection requiring systemic therapy.
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment

  o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Occurence of immune-related colitis associated with ipilimumab/nivolumab treatment | 28 months
  Occurence of grade 3 or higher immune-related colitis from the start of treatment with ipilimumab and nivolumab to 120 days after completion of treatment. Colitis will be graded using the Common Toxicity Criteria for Adverse Events version 4.02.

SECONDARY OUTCOMES:
Incidence of any immune-related adverse event associated with ipilimumab/nivolumab treatment | 28 months
  Incidence of any immune-related adverse event grade 3 or higher from the start of treatment with ipilimumab and nivolumab to 120 days after completion of treatment. Adverse events will be graded using the Common Toxicity Criteria for Adverse Events version 4.02.
Proportion of patients who discontinue treatment because of immune-related adverse events | 28 months
  Measured from the start of treatment with ipilimumab and nivolumab to 120 days after completion of treatment.
Objective response rate | Approximately 9 years (end of study)
  Objective response rate is defined as the proportion of patients achieving a complete response (disappearance of all lesions) and a partial response (30% or more decrease in the sum diameters of the target lesions) (Eisenhauer et al., 2009). Objective response rate will be measured using RECIST criteria version 1.1.
Changes in patient microbiome following FMT | At baseline (prior to FMT) and prior to the 1st, 2nd, 3rd and fourth dose of immunotherapy (approximately 1 week, 3 weeks, 7 weeks , and 10 weeks post FMT).
  Changes in patient microbiome will be determined by analysis of gut bacterial composition in patient stool samples at baseline and post-FMT.
Success rate of the fecal microbiota transplant | At baseline (prior to FMT) and prior to the 1st, 2nd, 3rd and fourth dose of immunotherapy (approximately 1 week, 3 weeks, 7 weeks , and 10 weeks post FMT).
  Success will be determined by comparing the make-up of the healthy donor microbiome to the patient's microbiome, using stool samples.
Determine the effect on immune response | At baseline (prior to FMT) and prior to the 1st, 2nd, 3rd and fourth dose of immunotherapy (approximately 1 week, 3 weeks, 7 weeks , and 10 weeks post FMT).
  Effects on the patient immune response will be assessed by examining changes in peripheral blood immune cells, chemokines, cytokines, and other immune and tumor biomarkers.
Health related quality of life | 30 months
  Patient reported quality of life will be measured using the standardized questionnaire, European Organization for Research and Treatment of Cancer (EORTC) EQ-5D-5L.

OTHER OUTCOMES:
Progression-free survival | Approximately 7 years
  The time from registration to death from any cause, or first recurrence of tumor at any site.
Overall survival | Approximately 7 years
  The time from registration to the time of death from any cause.
Assess the immune profile of the tumor | At baseline (prior to FMT) and between weeks 7 and 10.
  Tumor tissue will be collected at various timepoints, and will be used to examine the immune profile and changes of various genes in the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fernandes, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Saman Maleki, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Derived] Fernandes R, Jabbarizadeh B, Rajeh A, Hong MMY, Baines KJ, Ernst S, Winquist E, Ali AS, Penny S, Figueredo R, Parvathy SN, Lenehan JG, Pinto DM, Silverman MS, Maleki Vareki S. Fecal microbiota transplantation plus immunotherapy in metastatic renal cell carcinoma: the phase 1 PERFORM trial. Nat Med. 2026 Jan 28. doi: 10.1038/s41591-025-04183-8. Online ahead of print. PMID 41606120
- [Derived] Ninkov M, Schmerk CL, Moradizadeh M, Parvathy SN, Figueredo R, Burton JP, Silverman MS, Fernandes R, Maleki Vareki S, Haeryfar SMM. Improved MAIT cell functions following fecal microbiota transplantation for metastatic renal cell carcinoma. Cancer Immunol Immunother. 2023 May;72(5):1247-1260. doi: 10.1007/s00262-022-03329-8. Epub 2022 Nov 18. PMID 36396738